CLINICAL TRIAL: NCT00915382
Title: Phase III Trial of 3-weekly vs. 5-weekly Schedule of S-1 Plus Cisplatin Combination Chemotherapy for First Line Treatment of Advanced Gastric Cancer.
Brief Title: Trial of 3-weekly Versus 5-weekly Schedule of S-1 Plus Cisplatin in Gastric Cancer: SOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Kyungpook National University Hospital (Other); Seoul Veterans Hospital (Other); National Cancer Center, Korea (Other Government); Ulsan University Hospital (Other); Inje University (Other); Chonbuk National University Hospital (Other); Gachon University Gil Medical Center (Other); Korea Cancer Center Hospital (Other); Yeungnam University College of Medicine (Other); Hallym University Medical Center (Other); Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC0902
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — S 1 (combination); Cisplatin; titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3 weekly regimen of S-1 and cisplatin (Active Comparator)
  Interventions: Drug: S-1 and cisplatin
- 5 weekly regimen of S-1 and cisplatin (Active Comparator)
  Interventions: Drug: S-1 and cisplatin

INTERVENTIONS:
Drug: S-1 and cisplatin — S-1: 80 mg/m2/day po on Days 1-14
  cisplatin: 60 mg/m2 iv on Day 1
  Other Names: TS-1 and cisplatin
  Arms: 3 weekly regimen of S-1 and cisplatin
Drug: S-1 and cisplatin — S-1: 80 mg/day with BSA less than 1.25 m2, 100 mg/day with BSA more than 1.25 m2 and less than 1.5 m2, 120 mg/day with BSA more than 1.5 m2 on Days 1-21 and
  cisplatin: 60 mg/m2 iv on Day 1 or 8
  Other Names: TS-1 and cisplatin
  Arms: 5 weekly regimen of S-1 and cisplatin

SUMMARY:
The urgent need for a new effective therapy with better safety profile for the metastatic gastric cancer patients and promising results observed so far in the studies with S-1 plus cisplatin combination in advanced gastric cancer (AGC) strongly warrants the comparison of a 3-weekly schedule to a 5-weekly schedule of S-1 plus cisplatin as a standard regimen in the first-line treatment for AGC patients.

The objectives of this study are to compare a 3-weekly schedule to a 5-weekly schedule of S-1 plus Cisplatin combination in terms of efficacy, quality of life and safety in patients with previously untreated advanced or recurrent unresectable gastric cancer. Primary endpoint is progression-free survival. This is an open label, randomized, multi-center, non-inferiority/superiority (of 3-weekly regimen over 3-weekly regimen) hybrid study.

DETAILED DESCRIPTION:
The primary endpoint of this study is Progression Free Survival (PFS). It is defined as the time from the date of randomization to the time of disease progression as assessed by the investigators, or death due to any cause. The primary goal of this study is to compare two different schedules of S-1 plus cisplatin combination treatments (3-weekly regimen vs. 5-weekly regimen) for advanced gastric cancer with respect to the PFS based on the hybrid design where we can test superiority and non-inferiority in the same trial (Reference: Journal of Clinical Oncology 25: 5019-5023, 2007, Boris Freidlin, et el). First, the non-inferiority hypothesis will be tested based on the non-inferiority margin 1.15. If the inferiority cannot be rejected(meaning non-inferiority is proven) then the superiority will be tested. If the superiority test is positive, then superiority is concluded; otherwise non-inferiority without superiority will be concluded.

The sample size was calculated from the following consideration:

For non-inferiority test: non-inferiority margin 1.15, 10 percent reduction of hazard ratio, power 80 percent, alpha 0.025, accrual period 36 months, follow-up period 12 months, and the expected median PFS of 6 months for 5 weekly regimen were assumed. Based on the above considerations, total of 560 patients will be need. With 10 percent follow-up loss, we need 622 patients.

For superiority test: the median PFS for 5-weekly regimen is expected to be 6 months and 7.5 months for 3-weekly regimen. With sample size of 560 patients calculated above, for detecting 1.5 months difference in the median PFS between the two groups , we will have 81 percent of power, one-sided 5 percent type I error. Using the log rank test assuming exponential underlying distribution, accrual period of 36 months, minimum of 12 months follow-up after the last enrolment, 516 events will be needed to show the superiority of 3 week cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic or recurrent gastric adenocarcinoma including adenocarcinoma of the gastro-esophageal junction
* Age 18 to 74 years old
* Performance status (ECOG scale) 0-2
* No significant problems for oral intake and drug administration
* At least one measurable or evaluable disease defined by RECIST
* Adequate bone marrow function (ANC ≥ 1,500/uL, Platelet ≥ 100,000/ uL, Hb ≥ 9.0 g/dl)
* Adequate renal function: serum creatinine ≤ UNL (if serum creatinine > UNL, creatinine clearance should be ≥ 60 mL/min)
* Adequate hepatic function (Total bilirubin < 2 x UNL and AST/ALT levels < 3 x UNL without liver metastasis,total bilirubin < 3x ULN and AST/ALT levels < 5 x UNL with liver metastasis)
* Prior systemic therapy (for instance, cytotoxic chemotherapy or active/passive immunotherapy) is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study) and cisplatin was not used before
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Tumor type other than adenocarcinoma
* Previously exposed to any fluropymidine within 6 months before the study
* Previously exposed to Platinum therapy regardless of its period and/or duration
* Microscopic residual disease only after noncurative gastrectomy with R1 resection (resection margin positive)
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence)
* Prior radiotherapy was administered to target lesions selected for this study, or radiotherapy to the non-target lesions has been completed within 4 weeks before randomization
* Presence of CNS metastasis
* Major surgery within 4 weeks before initiation of study treatment or lack of complete recovery from the effects of major surgery (patient received curative operation or RFA for metastatic disease)
* Serious illness or medical conditions:

  * Congestive heart failure (NYHA class III or IV)
  * Unstable angina or myocardial infarction within the past 12 months
  * Significant arrhythmias requiring medication and conduction abnormality such as over 2nd degree AV block
  * Uncontrolled hypertension
  * Hepatic cirrhosis (≥ Child class B)
  * Interstitial pneumonia
  * Pulmonary adenomatosis
  * Psychiatric disorder that may interfere with protocol compliance
  * Unstable diabetes mellitus
  * Uncontrolled ascites or pleural effusion
  * Active infection
* Receiving a concomitant treatment interacting with S-1 or cisplatin:

  * Flucytosine (a fluorinated pyrimidine antifungal agent)
  * Antivirals such as sorivudine, ramivudine, brivudine or other chemically related agents, warfarin, phenprocoumon, phenytoin, allopurinol
* Pregnant or lactating woman
* Women of child bearing potential not using a contraceptive method
* Sexually active fertile men not using effective birth control during medication of study drug and up to 6 months after completion of study drug if their partners are women of child-bearing potential
* Any patients judged by the investigator to be unfit to participate in the study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2009-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
progression-free survival | accrual of patients for 36 months, followup of the last patient for 12 months

SECONDARY OUTCOMES:
overall survival | accrual of patients for 36 months, followup of the last patient for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center, Seoul, Korea; Won Ki Kang, M.D.PhD., Principal Investigator — Samsung Medical Center, Seoul, Korea; Jong Kwang Kim, M.D.PhD, Principal Investigator — Kyungpook National University Hospital, Korea; Young Iee Park, M.D.PhD, Principal Investigator — National Cancer Center, Korea; Jin Ho Baek, M.D.PhD., Principal Investigator — Ulsan University Hospital, Korea; Chang Hak Sohn, M.D.PhD., Principal Investigator — Inje University Pusan Paik Hospital, Korea; Eun Ki Song, M.D.PhD., Principal Investigator — Chonbuk National University Hospital, Korea; Dong Bok Shin, M.D.PhD., Principal Investigator — Gachon University Gil Medical Center; Sung Hyun Yang, M.D.PhD., Principal Investigator — Korea Cancer Center Hospital; Kyung Hee Lee, M.D.PhD., Principal Investigator — Yeungnam University College of Medicine; Dae Young Zang, M.D.PhD, Principal Investigator — Hallym University Medical Center; Ik-Joo Chung, M.D.PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Department of Oncology, Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Ryu MH, Baba E, Lee KH, Park YI, Boku N, Hyodo I, Nam BH, Esaki T, Yoo C, Ryoo BY, Song EK, Cho SH, Kang WK, Yang SH, Zang DY, Shin DB, Park SR, Shinozaki K, Takano T, Kang YK; SOS study investigators. Comparison of two different S-1 plus cisplatin dosing schedules as first-line chemotherapy for metastatic and/or recurrent gastric cancer: a multicenter, randomized phase III trial (SOS). Ann Oncol. 2015 Oct;26(10):2097-101. doi: 10.1093/annonc/mdv316. Epub 2015 Jul 27. PMID 26216386